CLINICAL TRIAL: NCT05334186
Title: Feasibility and Effectiveness of a Telehealth-Delivered Inductive Reasoning Training Program for Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB202101691
Record Dates: First submitted 2022-03-10; First posted 2022-04-19 (Actual); Last update posted 2022-10-21 (Actual); Status verified 2022-10

CONDITIONS: Reasoning Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Telehealth Reasoning Training (Experimental): Telehealth-delivered inductive reasoning training will focus on improving the ability to solve problems that require linear thinking and that follow a serial pattern or sequence. Participants will be taught strategies to identify patterns to solve problems. These problems involve identifying the pattern in series of numbers and letters, or recognizing patterns in everyday activities, like dosing for medications. Training will consist of ten training sessions, over 5 weeks, and will be conducted over Zoom. Each training session is 60-75 minutes long and typically consists of (a) 10 minutes of introductory training exercises for basic mental abilities, such as finding patterns in schedules, (b) training exercises for everyday tasks, such as filling out medication charts, recycling charts, and understanding medicine bottle labels, and (c) a 20-question practice assessment.
  Interventions: Behavioral: Telehealth Reasoning Training

INTERVENTIONS:
Behavioral: Telehealth Reasoning Training — The current study is explores the feasibility and preliminary relative effectiveness of a telehealth-delivered inductive reasoning intervention. The results of the study can help to provide insight on whether a telehealth-adapted reasoning training shows promise with older adults and can also be used to power future clinical trial studies to more definitively evaluate the effectiveness of telehealth delivered training.

SUMMARY:
This study seeks to investigate 1) whether telehealth-delivered cognitive training in reasoning, adapted from the in-person reasoning training program from the Advanced Cognitive Training for Independent and Vital Elderly (ACTIVE) clinical trial, is perceived well by older adult participants and therefore potentially feasible for future larger studies, and 2) whether the older adult participants improve as a function of telehealth-delivered reasoning training. More specifically, it proposes to investigate participants' perceptions of and compliance with a telehealth-delivered cognitive training intervention in reasoning and whether that intervention is effective in improving reasoning compared to ACTIVE's traditional face-to-face training and no-contact control groups. Innovations of the proposed study are: (a) to provide important insight into the participants' perceptions of and compliance with a telehealth-based cognitive training intervention in reasoning for older adults that could potentially be adapted in the future for clinical settings, and (b) to shed light on the relative effectiveness of telehealth-based cognitive training in reasoning.

DETAILED DESCRIPTION:
The proposed study is a pre-test post-test design exploring the feasibility and effectiveness of a telehealth-delivered inductive reasoning training program. The current study converts the widely disseminated in-person inductive reasoning training program from a large multisite clinical trial (ACTIVE) to a telehealth-delivered format. This study also benefits from the ability to compare telehealth delivered training to two propensity-matched comparison groups drawn from the ACTIVE sample of 2,802 adults aged 65 and older. The current study addresses whether telehealth-delivered training can achieve inductive reasoning improvements in older adults. In addition, because the delivery of the training is novel, and important aspect of this study is to assess how telehealth-delivered cognitive training in inductive reasoning is evaluated by older adult participants in terms of usefulness, ease of use & learnability, interface quality, interaction quality, reliability, and satisfaction/anticipated future use of the telehealth intervention.

ELIGIBILITY:
Inclusion Criteria:

* 65 years of age or older; have computer and internet; and are available during the duration of the study.

Exclusion Criteria:

* 64 years of age or younger
* Score < or = 22 on the Mini-Mental State Examination; have a diagnosis of Alzheimer's disease
* Have already experienced substantial functional decline (self-reported need for weight-bearing support or full caregiver performance of dressing, personal hygiene, or bathing 3 or more times in the previous 7 days)
* Have medical conditions that would predispose them to imminent functional decline or death (e.g., stroke within the past 12 months, certain cancers, or current chemotherapy or radiation treatment for cancer)
* Have recent cognitive training
* Are unavailable during the testing and intervention phases of the study
* Have severe losses in vision (self-reported difficulty in reading newsprint, or measured vision worse than 20/70 with best correction), hearing (interviewer-rated), or communicative ability (interviewer-rated) that would sufficiently impair performance to make participation impossible.
* Participants will also be excluded if they do not meet the criteria for telehealth readiness (being able to use Zoom and Canvas [an e-learning platform]).

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 34 (Actual)
Dates: Start 2022-02-25 (Actual); Primary Completion 2022-07-26 (Actual); Study Completion 2022-07-26 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Reasoning Performance to Post-Training Reasoning Performance: "Word Series" Measure | This will be administered 1 day to 21 days prior to reasoning training starting and after the ten sessions of inductive reasoning training are conducted, during the post-training assessment, which is 1-21 days after the final (tenth) training session.
  Word Series is a measure of reasoning, assessing what word would come next in a series.
Telehealth -Usability Questionnaire | This will be administered after the ten sessions of inductive reasoning training are conducted, during the post-training assessment, which is 1-21 days after the final (tenth) training session.
  A questionnaire assessing telehealth satisfaction. Answer choices range from Strongly Disagree, Disagree, Neutral, Agree, Strongly Agree. Higher scores = higher telehealth satisfaction.
Change from Baseline Reasoning Performance to Post-Training Reasoning Performance: "Letter Series" Measure | This will be administered 1 day to 21 days prior to reasoning training starting and after the ten sessions of inductive reasoning training are conducted, during the post-training assessment, which is 1-21 days after the final (tenth) training session.
  Letter Series is a measure of reasoning, assessing what letter would come next in a series.
Change from Baseline Reasoning Performance to Post-Training Reasoning Performance: "Letter Sets" Measure | This will be administered 1 day to 21 days prior to reasoning training starting and after the ten sessions of inductive reasoning training are conducted, during the post-training assessment, which is 1-21 days after the final (tenth) training session.
  Letter Sets is a measure of reasoning, assessing what set of letters is different from all the other sets of letters.

SECONDARY OUTCOMES:
Change from Baseline Vocabulary Performance to Post-Training Vocabulary Performance: "Vocabulary" Measure | This will be administered 1 day to 21 days prior to reasoning training starting and after the ten sessions of inductive reasoning training are conducted, during the post-training assessment, which is 1-21 days after the final (tenth) training session.
  The Vocabulary Measure is a measure of knowledge of word meanings.
Change from Baseline self-rated Health to Post-Training self-rated Health: "36-Item Short Form Survey (SF-36)" Measure | This will be administered 1 day to 21 days prior to reasoning training starting and after the ten sessions of inductive reasoning training are conducted, during the post-training assessment, which is 1-21 days after the final (tenth) training session.
  A questionnaire regarding self-rated health. Answer choices vary across questions.
Change from Baseline Personality in Intellectual-Aging Contexts to Post-Training Personality in Intellectual-Aging Contexts: "Personality in Intellectual-Aging Contexts" Questionnaire. | This will be administered 1 day to 21 days prior to reasoning training starting and after the ten sessions of inductive reasoning training are conducted, during the post-training assessment, which is 1-21 days after the final (tenth) training session.
  A questionnaire regarding Personality in Intellectual-Aging Contexts. Answer choice range from Strongly Disagree, Disagree, Slightly Disagree, Neutral, Slightly Agree, Agree, Strongly Agree.

CONTACTS AND LOCATIONS:
Overall Officials: Brad Taylor, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States